CLINICAL TRIAL: NCT01881113
Title: A Multi-Center, Double-Masked, Randomized, Vehicle-Controlled, Evaluation of the Onset and Duration of Action of AC-170 0.24% Ophthalmic Solution (Formula AFH-002) Compared to Vehicle (Formula AFH-001) in the Conjunctival Allergen Challenge (CAC) Model of Acute Allergic Conjunctivitis
Brief Title: A Multi-Center, Evaluation of the Onset and Duration of Action of AC-170 0.24% Compared to Vehicle
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aciex Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-100-0002
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Results first posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-10

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AC-170 0.24% (Experimental)
  Interventions: Drug: AC-170 0.24%
- AC-170 0% (Placebo Comparator)
  Interventions: Drug: AC-170 0%

INTERVENTIONS:
Drug: AC-170 0.24% — 1 drop in each eye at 2 separate times during a 14 day period
  Arms: AC-170 0.24%
Drug: AC-170 0% — 1 drop in each eye at 2 separate times during a 14 day period
  Arms: AC-170 0%

SUMMARY:
The purpose of this study is to evaluate the onset and duration of action of AC-170 0.24% compared to vehicle in the prevention of the signs and symptoms of allergic conjunctivitis in the conjunctival allergen challenge (CAC) model.

ELIGIBILITY:
Inclusion Criteria:

* positive bilateral conjunctival allergen challenge (CAC) reaction

Exclusion Criteria:

* known contraindications or sensitivities to the study medication or its components
* any ocular condition that, in the opinion of the investigator, could affect the subjects safety trial parameters
* use of disallowed medication during the period indicated prior to the enrollment or during the study

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene McLaurin, MD, Principal Investigator — Total Eye Care, PA; Edward Meier, MD, Principal Investigator — Eye Care Associates of Greater Cincinnati; Mark Bergmann, MD, Principal Investigator — Eye Care Associates of Greater Cincinnati
Locations (1):
- Ora, Inc., Andover, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from three sites in the US.
Pre-assignment Details: There were 101 subjects enrolled, 14 subjects discontinued, and 87 subjects completed the study. Participant flow and baseline characteristics are presented for the 101 subjects that met all inclusion criteria and none of the exclusion criteria and were randomized to receive AC-170 0.24% or Vehicle.
Period: Overall Study
Arm/Group | AC-170 0.24% | AC-170 0%
Started | 51 | 50
Completed | 43 | 44
Not Completed | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AC-170 0.24% | AC-170 0% | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (12.8) | 39.2 (10.84) | 39.9 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 20 | 32
  Male | 39 | 30 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 50 | 50 | 100
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 17 | 27
  White | 41 | 31 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 51 | 50 | 101

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching at Duration of Action (8 Hours + 30 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 8 hours + 30 minutes after drop instillation. Ocular itching was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ocular itching score over both eyes was analyzed.
Time Frame: 3, 5, 7 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 51 | 50
units on a scale
  3 minutes post-CAC | 1.94 (0.933) | 2.86 (0.748)
  5 minutes post-CAC | 2.03 (0.947) | 2.94 (0.712)
  7 minutes post-CAC | 1.82 (1.026) | 2.66 (0.809)

2. Primary Outcome: Ocular Itching at Onset of Action (15 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Ocular itching was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ocular itching score over both eyes was analyzed.
Time Frame: 3, 5, 7 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 51 | 50
units on a scale
  3 minutes post-CAC | 1.01 (1.006) | 2.54 (0.943)
  5 minutes post-CAC | 1.17 (1.002) | 2.51 (0.875)
  7 minutes post-CAC | 1.15 (1.006) | 2.23 (0.956)

3. Primary Outcome: Conjunctival Redness at Duration of Action (8 Hours + 30 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 8 hours + 30 minutes after drop instillation. Conjunctival Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of conjunctival redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 51 | 50
units on a scale
  7 minutes post-CAC | 1.97 (0.702) | 2.39 (0.619)
  15 minutes post-CAC | 2.13 (0.639) | 2.38 (0.602)
  20 minutes post-CAC | 2.09 (0.701) | 2.40 (0.639)

4. Primary Outcome: Conjunctival Redness at Onset of Action (15 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Conjunctival Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of conjunctival redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 51 | 50
units on a scale
  7 minutes post-CAC | 1.92 (0.713) | 2.38 (0.653)
  15 minutes post-CAC | 2.19 (0.608) | 2.37 (0.661)
  20 minutes post-CAC | 2.15 (0.646) | 2.41 (0.651)

5. Secondary Outcome: Ciliary Redness at Duration of Action (8 Hours + 30 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 8 hours + 30 minutes after drop instillation. Ciliary Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ciliary redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT). Number of analyzed subjects differ due to subject discontinuation during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 50 | 48
units on a scale
  7 minutes post-CAC | 1.71 (0.794) | 2.15 (0.689)
  15 minutes post-CAC | 1.93 (0.753) | 2.05 (0.777)
  20 minutes post-CAC | 1.87 (0.801) | 2.19 (0.659)

6. Secondary Outcome: Ciliary Redness at Onset of Action (15 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Ciliary Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ciliary redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT). Number of analyzed subjects differ due to subject discontinuation during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 43 | 44
units on a scale
  7 minutes post-CAC | 1.62 (0.945) | 2.29 (0.803)
  15 minutes post-CAC | 2.05 (0.793) | 2.34 (0.780)
  20 minutes post-CAC | 2.09 (0.779) | 2.36 (0.784)

7. Secondary Outcome: Episcleral Redness at Duration of Action (8 Hours + 30 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 8 hours + 30 minutes after drop instillation. Episcleral Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of episcleral redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT). Number of analyzed subjects differ due to subject discontinuation during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 50 | 48
units on a scale
  7 minutes post-CAC | 1.92 (0.662) | 2.29 (0.567)
  15 minutes post-CAC | 2.08 (0.663) | 2.27 (0.605)
  20 minutes post-CAC | 2.06 (0.689) | 2.30 (0.640)

8. Secondary Outcome: Episcleral Redness at Onset of Action (15 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Episcleral Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of episcleral redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT). Number of analyzed subjects differ due to subject discontinuation during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 43 | 44
units on a scale
  7 minutes post-CAC | 1.91 (0.798) | 2.31 (0.575)
  15 minutes post-CAC | 2.22 (0.645) | 2.32 (0.582)
  20 minutes post-CAC | 2.18 (0.655) | 2.36 (0.604)

9. Secondary Outcome: Chemosis at Duration of Action (8 Hours + 30 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 8 hours + 30 minutes after drop instillation. Chemosis was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of chemosis score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT). Number of analyzed subjects differ due to subject discontinuation during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 50 | 48
units on a scale
  7 minutes post-CAC | 0.63 (0.540) | 0.96 (0.666)
  15 minutes post-CAC | 0.89 (0.627) | 1.28 (0.773)
  20 minutes post-CAC | 0.95 (0.753) | 1.27 (0.785)

10. Secondary Outcome: Chemosis at Onset of Action (15 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Chemosis was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of chemosis score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT). Number of analyzed subjects differ due to subject discontinuation during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 43 | 44
units on a scale
  7 minutes post-CAC | 0.35 (0.387) | 0.58 (0.519)
  15 minutes post-CAC | 0.59 (0.585) | 0.75 (0.671)
  20 minutes post-CAC | 0.67 (0.626) | 0.85 (0.702)

11. Secondary Outcome: Eyelid Swelling at Duration of Action (8 Hours + 30 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 8 hours + 30 minutes after drop instillation. Eyelid swelling was assessed by the patient on a 0-3 scale (0=none to 3=severe). Average of eyelid swelling score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT). Number of analyzed subjects differ due to subject discontinuation during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 50 | 48
units on a scale
  7 minutes post-CAC | 0.7 (0.70) | 1.4 (0.78)
  15 minutes post-CAC | 0.8 (0.71) | 1.4 (0.80)
  20 minutes post-CAC | 0.9 (0.91) | 1.4 (0.89)

12. Secondary Outcome: Eyelid Swelling at Onset of Action (15 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Eyelid swelling was assessed by the patient on a 0-3 scale (0=none to 3=severe). Average of eyelid swelling score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT). Number of analyzed subjects differ due to subject discontinuation during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 43 | 44
units on a scale
  7 minutes post-CAC | 0.4 (0.67) | 1.2 (0.63)
  15 minutes post-CAC | 0.5 (0.76) | 1.3 (0.75)
  20 minutes post-CAC | 0.4 (0.70) | 1.2 (0.77)

13. Secondary Outcome: Tearing at Duration of Action (8 Hours + 30 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 8 hours + 30 minutes after drop instillation. Tearing was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of tearing score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT). Number of analyzed subjects differ due to subject discontinuation during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 50 | 48
units on a scale
  7 minutes post-CAC | 0.8 (0.67) | 1.2 (0.81)
  15 minutes post-CAC | 0.8 (0.90) | 1.2 (0.94)
  20 minutes post-CAC | 0.9 (0.98) | 1.0 (1.01)

14. Secondary Outcome: Tearing at Onset of Action (15 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Tearing was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of tearing score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT). Number of analyzed subjects differ due to subject discontinuation during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 43 | 44
units on a scale
  7 minutes post-CAC | 0.5 (0.61) | 1.1 (0.89)
  15 minutes post-CAC | 0.5 (0.62) | 1.1 (0.90)
  20 minutes post-CAC | 0.5 (0.65) | 1.0 (0.94)

15. Secondary Outcome: Rhinorrhea at Duration of Action (8 Hours + 30 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 8 hours + 30 minutes after drop instillation. Rhinorrhea was assessed by the patient on a 0-4 scale (0=none to 4=severe). Rhinorrhea score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT). Number of analyzed subjects differ due to subject discontinuation during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 50 | 48
units on a scale
  7 minutes post-CAC | 0.6 (0.85) | 1.1 (0.88)
  15 minutes post-CAC | 0.8 (0.89) | 1.3 (1.00)
  20 minutes post-CAC | 1.0 (1.01) | 1.3 (1.06)

16. Secondary Outcome: Rhinorrhea at Onset of Action (15 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Rhinorrhea was assessed by the patient on a 0-4 scale (0=none to 4=severe). Rhinorrhea score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT). Number of analyzed subjects differ due to subject discontinuation during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 43 | 44
units on a scale
  7 minutes post-CAC | 0.5 (0.70) | 1.3 (1.05)
  15 minutes post-CAC | 0.7 (0.89) | 1.3 (1.12)
  20 minutes post-CAC | 0.8 (0.78) | 1.1 (1.05)

17. Secondary Outcome: Nasal Pruritus at Duration of Action (8 Hours + 30 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 8 hours + 30 minutes after drop instillation. Nasal Pruritus was assessed by the patient on a 0-4 scale (0=none to 4=severe). Nasal Pruritus score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT). Number of analyzed subjects differ due to subject discontinuation during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 50 | 48
units on a scale
  7 minutes post-CAC | 0.5 (0.79) | 0.9 (0.99)
  15 minutes post-CAC | 1.0 (1.01) | 1.0 (1.11)
  20 minutes post-CAC | 0.9 (1.00) | 0.9 (0.96)

18. Secondary Outcome: Nasal Pruritus at Onset of Action (15 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Nasal Pruritus was assessed by the patient on a 0-4 scale (0=none to 4=severe). Nasal Pruritus score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT). Number of analyzed subjects differ due to subject discontinuation during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 43 | 44
units on a scale
  7 minutes post-CAC | 0.4 (0.76) | 0.8 (0.87)
  15 minutes post-CAC | 0.6 (1.05) | 0.8 (0.99)
  20 minutes post-CAC | 0.6 (0.87) | 0.9 (0.95)

19. Secondary Outcome: Ear or Palate Pruritus at Duration of Action (8 Hours + 30 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 8 hours + 30 minutes after drop instillation. Ear or Palate Pruritus was assessed by the patient on a single 0-4 scale (0=none to 4=severe). Ear or Palate Pruritus score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT). Number of analyzed subjects differ due to subject discontinuation during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 50 | 48
units on a scale
  7 minutes post-CAC | 0.4 (0.73) | 1.2 (1.10)
  15 minutes post-CAC | 0.8 (1.00) | 1.5 (1.25)
  20 minutes post-CAC | 1.0 (1.14) | 1.6 (1.27)

20. Secondary Outcome: Ear or Palate Pruritus at Onset of Action (15 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Ear or Palate Pruritus was assessed by the patient on a single 0-4 scale (0=none to 4=severe). Ear or Palate Pruritus score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT). Number of analyzed subjects differ due to subject discontinuation during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 43 | 44
units on a scale
  7 minutes post-CAC | 0.3 (0.74) | 0.8 (0.96)
  15 minutes post-CAC | 0.6 (1.05) | 1.3 (1.17)
  20 minutes post-CAC | 0.7 (1.06) | 1.3 (1.24)

21. Secondary Outcome: Nasal Congestion at Duration of Action (8 Hours + 30 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 8 hours + 30 minutes after drop instillation. Nasal Congestion was assessed by the patient on a 0-4 scale (0=none to 4=severe). Nasal Congestion score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT). Number of analyzed subjects differ due to subject discontinuation during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 50 | 48
units on a scale
  7 minutes post-CAC | 0.5 (0.68) | 1.0 (0.89)
  15 minutes post-CAC | 0.8 (0.85) | 1.4 (1.08)
  20 minutes post-CAC | 1.1 (1.08) | 1.3 (1.00)

22. Secondary Outcome: Nasal Congestion at Onset of Action (15 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Nasal Congestion was assessed by the patient on a 0-4 scale (0=none to 4=severe). Nasal Congestion score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT). Number of analyzed subjects differ due to subject discontinuation during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 43 | 44
units on a scale
  7 minutes post-CAC | 0.4 (0.73) | 1.1 (1.13)
  15 minutes post-CAC | 0.5 (0.86) | 1.3 (1.17)
  20 minutes post-CAC | 0.6 (0.85) | 1.3 (1.14)

23. Secondary Outcome: Percentage of Participants With At Least One Nasal Symptom at Duration of Action (8 Hours + 30 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 8 hours + 30 minutes after drop instillation. For Nasal Composite Score the Total Composite Score ranges from 0 to 16, higher scores represent greater severity. Patients needed to have at least one of the nasal symptoms present (Rhinorrhea + Nasal Pruritus + Ear or Palate Pruritus + Nasal Congestion) each symptom was assessed by the patient on a 0-4 scale (0=none to 4=severe). Nasal Composite score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT). Number of analyzed subjects differ due to subject discontinuation during the study.
Measure: Number; unit: % of participants
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 50 | 48
% of participants
  7 minutes post-CAC | 58 | 87.5
  15 minutes post-CAC | 78 | 89.6
  20 minutes post-CAC | 84 | 89.6

24. Secondary Outcome: Percentage of Participants With At Least One Nasal Symptom at Onset of Action (15 Minutes Post-Dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. For Nasal Composite Score the Total Composite Score ranges from 0 to 16, higher scores represent greater severity. Patients needed to have at least one of the nasal symptoms present (Rhinorrhea + Nasal Pruritus + Ear or Palate Pruritus + Nasal Congestion) each symptom was assessed by the patient on a 0-4 scale (0=none to 4=severe). Nasal Composite score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT). Number of analyzed subjects differ due to subject discontinuation during the study.
Measure: Number; unit: % of participants
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 43 | 44
% of participants
  7 minutes post-CAC | 51.2 | 81.8
  15 minutes post-CAC | 58.1 | 86.4
  20 minutes post-CAC | 72.1 | 88.6

25. Secondary Outcome: Tolerability of Study Medication at Visit 3A
Description: Tolerability was assessed upon instillation of study medication, at 1 minute and 2 minutes post study medication instillation. Drop comfort was assessed using a 0-to 10 scale where 0=very comfortable and 10=very uncomfortable.
Time Frame: upon instillation, 1 minute and 2 minutes post instillation
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-170 0.24% | AC-170 0%
Number analyzed (Participants) | 51 | 50
units on a scale
  Upon instillation | 1.6 (2.02) | 0.8 (1.22)
  1 minute post-instillation | 3.0 (2.33) | 1.1 (1.14)
  2 minutes post-instillation | 2.6 (2.14) | 1.1 (1.13)

ADVERSE EVENTS:
Time Frame: Adverse events were collected through study completion, an average of 5 weeks.. All subjects who received study medication were evaluable for the safety analysis.
Description: Throughout the visits, staff collected all Adverse Events reported, elicited, or observed.
Arm/Group | AC-170 0.24% | AC-170 0%
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/50
Other Adverse Events (participants affected / at risk) | 3/51 | 5/50
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AC-170 0.24% (N=51) | AC-170 0% (N=50)
Visual acuity reduced (Eye disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes